CLINICAL TRIAL: NCT01434212
Title: Study of Parameters of Early Hepatitis C Virus Dynamics for Predicting the Outcome of Standard Interferon Therapy With Chinese Cohort
Brief Title: Patterns of Early Hepatitis C Virus Decline Predict the Outcome of Interferon Therapy
Acronym: sIFN-pred1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Junqi Niu, Vice-President of First Hospital of Jilin University, The First Hospital of Jilin University
Other Study IDs: 2008ZX10004-002-jida01; 2008ZX10002-014-jida01 (Other: China: Ministry of Science and Technology); 2009ZX10004-105-jida01 (Other: China: Ministry of Science and Technology)
Record Dates: First submitted 2011-09-08; First posted 2011-09-14 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Hepatitis
Keywords: HCV dynamics; Mathematical model; Interferon; Predict; Hepatitis C Virus
MeSH Terms: conditions — Hepatitis; Hepatitis C | interventions — Interferon alpha-2; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum,Peripheral blood mononuclear cells (PBMC)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Interferon and ribavirin: All the patients followed the standard treatment protocol.
  Interventions: Drug: Interferon Alfa-2b, Ribavirin

INTERVENTIONS:
Drug: Interferon Alfa-2b, Ribavirin — Interferon:dosage,5 million units/person;frequency,every other day (qod);duration,48 weeks;Subcutaneous injection.
  Ribavirin: dosage,15mg/kg/day;frequency,three times a day (t.i.d);duration,48 weeks;take orally.
  Other Names: Generic: Recombinant Human Interferon alpha-2b,Ribavirin; Brand: Kaiyinyisheng,Weilake; FDA Approval number:S20030032,H10940157

SUMMARY:
The purpose of this study is to determine whether the outcome of interferon therapy on HCV infected patients can be early precisely predicted with a novel mathematic method with Chinese population.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection rate in China is about 3%, which means about 30 million patients. Combination therapy of ribavirin and interferons (IFN) is the standard clinical treatment of HCV chronical infections. However, overall rate of sustained virological response (SVR) still do not exceed 60% even with ribavirin and peg-IFN. Due to several virus- and patient-related factors, treatment is even less successful in certain populations, especially in HCV genotype 1 infection. Thus the standard therapy duration is optimized according to the virus genotype in the clinical practice. Nowadays, two direct antiviral agents (DAAs) have been approved by Food and Drug Administration (FDA) of USA this year, which increases the SVR rate. However, high price, side effects and long duration render people to hesitate about the addition of the third drug in the traditional prescription.

Predicting the outcome of traditional therapy is the cornerstone of the personalized therapy for HCV infected patients. In order to obtain an accurate prediction, different methods have been tried. Several indicators have been suggested to predict the final treatment outcomes. Rapid Virus Response (RVR), which indicates the non-detectable virus at the forth week since therapy starts, has been used to predict the final treatment outcome.Other indicators, including virus genotype, host genotype of IL-28B, human race and interferon stimulated genes (ISG) expression have also been shown to relate to and be able to predict the treatment outcomes to some extent. Here the investigators propose that the HCV virus dynamics analysis will give a more precise prediction for the therapy outcome.

The general idea is that blood HCV titration data is obtained continuously in the early treatment period (first 6 weeks) of the patients who have strictly followed the therapy method. These titration data will be used to draw virus dynamics curve and calculate the corresponding parameters individually. The parameter(s) that can distinguish patients who reach the therapy evaluation standard from those who failed to reach the evaluation standard will be selected out, and such parameter(s) may be used to predict the therapy outcome of a new patient in the early stage of his/her treatment.

ELIGIBILITY:
Inclusion Criteria:

* Serologic evidence of chronic hepatitis C infection by an anti-HCV antibody test
* Serum HCV-RNA > 3 log IU/ml
* Has been infected by HCV for more than 6 months
* ALT,AST have been elevated continuously, inflammation and necrosis have been observed according to the histology diagnosis (G>=2),modest liver fibrosis (S>=2)
* For those patients whose ALT are normal,treatment accord to the liver biopsy. If obvious fibrosis has been detected (S2,S3),treatment should be done.For those S0,S1 stage patients, treatment could be delayed, but ALT/AST should be assayed every 3-6 months.
* Compensated liver disease
* Patients have never been treated with traditional interferon plus ribavirin or peginterferon plus ribavirin

Exclusion Criteria:

History:

* Has history of decompensated liver diseases
* Has been treated with other anti-virus drugs,or anti-tumor drugs,immuno-suppression drugs
* Has a history of autoimmune hepatitis
* History of a severe seizure disorder or current anticonvulsant use
* History or other evidence of a medical condition associated with chronic liver disease other than HCV which would make the patient, in the opinion of the investigator, unsuitable for the study (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4g/dL (as may be seen with ribavirin therapy) would not be well-tolerated
* History of thyroid disease poorly controlled on prescribed medications, elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease

Current condition:

* Pregnant women or women during the lactation period
* Co-infected with hepatitis b virus or human immunodeficiency virus
* Liver cancer or alpha-fetoprotein > 100ng/ml
* Blood neutrophils count < 1500/mm3, or platelets count < 90000/mm3
* Female hemoglobin <11.5g/dL, male hemoglobin <12.5g/dL
* Blood creatinine > 1.5 ULN
* Have severe mental diseases,especially depression
* Severe pulmonary dysfunction
* Severe cardiovascular disease
* Uncontrolled diabetes
* Uncontrolled thalassemia
* Evidence of alcohol abuse (alcohol consumption>40 g/day)
* Unwillingness to provide informed consent or abide by the requirements of the study
* Local or System malignancy unstable status

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are from the northeast of China. Most of the patients have been infected by the hepatitis c virus due to the drug abuse. Many of them share the same syringe for drug intravenous injection. However, HIV infection has been rarely detected.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Blood HCV RNA Copies | 0h,8h,10h,12h,18h,24h,37h,43h,3d,7d,2w,4w,6w,12w,24w,48w
  Blood HCV RNA copies were assayed with Roche - COBAS® AmpliPrep/COBAS® TaqMan® HCV Test.

SECONDARY OUTCOMES:
IL-28B polymorphism | Baseline
  IL28 gene polymorphism,rs8099917,rs12979860,etc
Microarray Analysis of PBMC Gene Expression | Baseline,8h,18h,3d
  During the first 3 days, blood samples are collected for PBMC separation and microarray analysis.
HCV genotype | Baseline
  HCV NS5A is cloned into T vector and sequenced for evolutionary analysis.
Blood Anti-HCV,HBV Antibody | Baseline
  Co-infection status are analyzed.
HCV genome sequencing | 0h,8h,10h,12h,18h,24h,37h,43h,3d
  Deep sequencing is used for blood serum HCV genome analysis.
Alanine Aminotransferase (ALT) and Aspartate transaminase (AST) | Baseline,4w,6w,12w,24w,48w
  ALT AST are assayed to detect the hepatic function.
Fibrosis stage | Baseline,4w,12w,24w,48w
  Fibrosis is analyzed with Fibroscan.
Regular blood test | Baseline,4w,12w,24w,48w
  The distribution and absolute count of the different types of blood cells are assayed.
Electrocardiography | Baseline,4w,12w,24w,48w
  Electrocardiography is taken to avoid severe side effects.
Alcohol ,smoking condition | Baseline,4w,12w,24w,48w
  Patients are asked whether they take alcohol or smoke cigarettes during the therapy period.
Drug abuse history | Baseline
  Patients will be asked about their drug usage history.

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, PhD/MD, Study Chair — First Hospital Jilin University; Bing Sun, PhD/MD, Principal Investigator — Chinese Academy of Sciences
Locations (1):
- First Hospital Jilin University, Changchun, Jilin, China

REFERENCES:
- [Background] Neumann AU, Lam NP, Dahari H, Gretch DR, Wiley TE, Layden TJ, Perelson AS. Hepatitis C viral dynamics in vivo and the antiviral efficacy of interferon-alpha therapy. Science. 1998 Oct 2;282(5386):103-7. doi: 10.1126/science.282.5386.103. PMID 9756471
- [Background] Dahari H, Ribeiro RM, Perelson AS. Triphasic decline of hepatitis C virus RNA during antiviral therapy. Hepatology. 2007 Jul;46(1):16-21. doi: 10.1002/hep.21657. PMID 17596864
- [Background] Snoeck E, Chanu P, Lavielle M, Jacqmin P, Jonsson EN, Jorga K, Goggin T, Grippo J, Jumbe NL, Frey N. A comprehensive hepatitis C viral kinetic model explaining cure. Clin Pharmacol Ther. 2010 Jun;87(6):706-13. doi: 10.1038/clpt.2010.35. Epub 2010 May 12. PMID 20463660
- [Background] Dixit NM, Layden-Almer JE, Layden TJ, Perelson AS. Modelling how ribavirin improves interferon response rates in hepatitis C virus infection. Nature. 2004 Dec 16;432(7019):922-4. doi: 10.1038/nature03153. PMID 15602565
- [Background] Manns MP, McHutchison JG, Gordon SC, Rustgi VK, Shiffman M, Reindollar R, Goodman ZD, Koury K, Ling M, Albrecht JK. Peginterferon alfa-2b plus ribavirin compared with interferon alfa-2b plus ribavirin for initial treatment of chronic hepatitis C: a randomised trial. Lancet. 2001 Sep 22;358(9286):958-65. doi: 10.1016/s0140-6736(01)06102-5. PMID 11583749
- [Background] Dill MT, Duong FH, Vogt JE, Bibert S, Bochud PY, Terracciano L, Papassotiropoulos A, Roth V, Heim MH. Interferon-induced gene expression is a stronger predictor of treatment response than IL28B genotype in patients with hepatitis C. Gastroenterology. 2011 Mar;140(3):1021-31. doi: 10.1053/j.gastro.2010.11.039. Epub 2010 Nov 25. PMID 21111740
- [Background] Araujo ES, Dahari H, Neumann AU, de Paula Cavalheiro N, Melo CE, de Melo ES, Layden TJ, Cotler SJ, Barone AA. Very early prediction of response to HCV treatment with PEG-IFN-alfa-2a and ribavirin in HIV/HCV-coinfected patients. J Viral Hepat. 2011 Apr;18(4):e52-60. doi: 10.1111/j.1365-2893.2010.01358.x. PMID 20738775